CLINICAL TRIAL: NCT03273400
Title: Investigating the Effect of L4 and L5 Lumbar Posterior -Anterior Mobilisations on Measures of Lumbar and Hamstring Range of Motion, and Electromyography Activity of the Erector Spinae and Hamstring
Brief Title: Effect of Mobilisations on Lumbar and Hamstring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Paul Chesterton, Senior Lecturer Sport and Exercise, Teesside University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TeessideU
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Hamstring Injury
Keywords: Lumbar, Hamstring, Mobilisation

STUDY DESIGN:
Intervention Model Description: The study will be a cross-over design. A pre-test post-test design will be used to evaluate the sEMG activity of the Erector Spinae muscle group and the Hamstring muscle (Biceps Femoris). Lumbar flexion range of motion and hamstring length will be tested prior too mobilisations and post intervention immediate and at intervals of 5, 10, 15, 20, 30, 60 minutes. Participants will be receive non-intervention one week and mobilisations the following week.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilisations (Experimental): The intervention will consist of unilateral lumbar mobilisations at the L4 and L5 level in a Posterior Anterior direction. The plinth will rest on force plates to allow the authors to analyse the force placed through the vertebrae. Grade three mobilisations will be applied for a one minute period three times at both L4 and L5 level. Each level will be determined by a passive physiological intervertebral movement. Participants will receive the mobilisations at L5 first for one minute followed by L4. This is an appropriate dose for mobilisation application (Maitland, 2013). This process will be carried out three times.
  Following the intervention all measure lumbar flexion, hamstring extensibility and sEMG activity will be recorded immediately, 5, 10, 15, 20, 30, 60 minutes post application as a single test.
  Interventions: Other: Lumbar Mobilisations
- Control (No Intervention): All outcome measures (lumbar/hamstring range of motion; EMG activity of the Biceps Femoris and Erector Spinae) will be measured. The control group will then receive no intervention and be asked to lie supine on a plinth for the treatment duration before having the outcome measures reassessed.

INTERVENTIONS:
Other: Lumbar Mobilisations — Please see arm (intervention) description
  Arms: Mobilisations

SUMMARY:
To compare the immediate and short-term effects of L4 and L5 Unilateral Posterior Anterior (UPA) Mobilisations on the lumbar and hamstring range of motion and EMG activity of the Erector Spinae and Hamstring muscles.

Using a pre-test post-test crossover design subjects lumbar flexion and active knee extension with be recorded prior to and following unilateral zygapophyseal joint mobilisations. Measures will be taken immediately after and then 5, 10, 15, 20, 30 and 60 minutes intervals post intervention. Mobilisation force will be measured via force plates to ensure consistent mobilisation pressure.

Following data collection statistical analysis will be undertaken to analyse any potential benefit of lumbar mobilisations to influence the EMG activity of the Erector Spinae and Hamstrings. Functional assessment of lumbar range of motion and hamstring range of motion to be conducted and analyse any effect on movement

DETAILED DESCRIPTION:
25-30 participants will be tested in the Olympia Building Biomechanics Laboratory at Teesside University.

Due to the nature of the cross-over design participants will attend the laboratory twice, one week apart.

Baseline measurements of Lumbar flexion and hamstring range of motions will be taken.

During lumbar flexion participants will be asked to stand with their arms at their side (anatomical position) and feet 8cm part. The tester will demonstrate the flexion motion then request the subject bends forwards are far as is possible, maintaining knee extension. A previous reliability study (Page 2012) has indicated four lumbar flexion movements repetitions were required to prevent the effects of passive stiffness improving the range. On the fourth trial the measurement via the modified schober test. This requires skin markers to be placed 10cm above and 5cm below the lumbar-sacral junction and the change distance calculated at end range. This will be conducted by the lead author, Paul Chesterton, a physiotherapist with appropriate insurance and qualifications.

Hamstring extensibility will be measured via the active knee extension test. Test leg will be determined by dominant/kicking leg. Subjects will be secured into anterior pelvic tilt via a belt and asked to extend the knee to maximal length. A purpose made wooden wedge will provide a right angle surface to ensure the hip is held at 90 degrees. The digital inclinometer will record the change in degrees of active knee extension post-test. The knee will be extended to end range, determined by the subject, with the hip, knee and ankle maintained in neutral. The non-dominant leg will be secured to the bed via a belt.

To record the surface electromyography (SEMG) activity in the muscles of the participants in this study the Zerowire Cometa system will be used. This system will record the muscle activity wirelessly. Every electrode unit is equipped with a small unit for signal processing and transmission to the data receiver. The electrodes are single use disposable, self-adhesive silver chloride dual snap on electrodes pre-set at a distance of 20mm.

All participants will have the skin prepared prior to the noraxon electrode being placed on their skin. Skin preparation will consist of shaving the area to remove any hair then wiping the area with alcohol wipe then the placing noraxon dual electrode in appropriate position in relation to recommendations by Seniam (2003). The electrodes are placed in line to the pennant of the muscle.

Electrodes will be attached according to European recommendation (seniam) at the Paraspinal muscles, and the Biceps Femoris of the dominant leg. A baseline sEMG will then be taken whilst the participant is at rest for 60seconds. The electrode placement and sEMG recording will be taken by a qualified laboratory technician employed by Teesside University.

The intervention will consist of unilateral lumbar mobilisations at the L4 and L5 level in a Posterior Anterior direction. The plinth will rest on force plates to allow the authors to analyse the force placed through the vertebrae. Grade three mobilisations will be applied for a one minute period three times at both L4 and L5 level. Each level will be determined by a passive physiological intervertebral movement. Participants will receive the mobilisations at L5 first for one minute followed by L4. This is an appropriate dose for mobilisation application (Maitland, 2013). This process will be carried out three times.

Following either the control or intervention all measure lumbar flexion, hamstring extensibility and sEMG activity will be recorded immediately, 5, 10, 15, 20, 30, 60 minutes post application as a single test.

Data analysis will occur using the zerowire cometa system version 1.6. The raw rate will be smoothed and rectified using a Butterworth algorithm with a high pass filter with a cut of frequency of 20Hz at order 5 with the data will be rectified using route mean square (RMS) set at a window of 20ms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65. Participants willing to provide inform consent. Participants who successfully complete the medical questionnaire. No current lower back or lower limb pathology.

Exclusion Criteria:

* Current symptomatic low back pain or lower limb pathology. Participants with altered neurodynamic symptoms. Previous lumbar surgery. Under supervision of another health practionare Pregnant participants Contraindications or precautions to spinal mobilisation

  * malignancy, inflammatory or infectious processes involving the spine or peripheral joints,
  * osteoporosis,
  * spinal disorders including spondylolisthesis, ankylosing spondylitis, spinal fusion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Lumbar Range of Motion | 5, 10, 15, 20, 30, 60 minutes post application as a single test.
  During lumbar flexion participants will be asked to stand with their arms at their side (anatomical position) and feet 8cm part. The tester will demonstrate the flexion motion then request the subject bends forwards are far as is possible, maintaining knee extension. A previous reliability study (Page 2012) has indicated four lumbar flexion movements repetitions were required to prevent the effects of passive stiffness improving the range. On the fourth trial the measurement via the modified schober test. This requires skin markers to be placed 10cm above and 5cm below the lumbar-sacral junction and the change distance calculated at end range.
Hamstring Range of Motion | 5, 10, 15, 20, 30, 60 minutes post application as a single test.
  Hamstring extensibility will be measured via the active knee extension test. Test leg will be determined by dominant/kicking leg. Subjects will be secured into anterior pelvic tilt via a belt and asked to extend the knee to maximal length. A purpose made wooden wedge will provide a right angle surface to ensure the hip is held at 90 degrees. The digital inclinometer will record the change in degrees of active knee extension post-test. The knee will be extended to end range, determined by the subject, with the hip, knee and ankle maintained in neutral. The non-dominant leg will be secured to the bed via a belt.
Electromyography of Erector Spinae | 5, 10, 15, 20, 30, 60 minutes post application as a single test.
  Record electromyography (SEMG) activity in the muscles of the participants in this study the Zerowire Cometa system will be used. Every electrode unit is equipped with a small unit for signal processing and transmission to the data receiver. The electrodes are single use disposable, self-adhesive silver chloride dual snap on electrodes pre-set at a distance of 20mm.
  All participants will have the skin prepared prior to the noraxon electrode being placed on their skin. Electrodes will be attached according to European recommendation (seniam) at the Paraspinal muscles (L1 region). A baseline sEMG will then be taken whilst the participant is at rest for 60seconds. The electrode placement and sEMG recording will be taken by a qualified laboratory technician employed by Teesside University.
Electromyography of Biceps Femoris | 5, 10, 15, 20, 30, 60 minutes post application as a single test.
  Record electromyography (SEMG) activity in the muscles of the participants in this study the Zerowire Cometa system will be used. Every electrode unit is equipped with a small unit for signal processing and transmission to the data receiver. The electrodes are single use disposable, self-adhesive silver chloride dual snap on electrodes pre-set at a distance of 20mm.
  All participants will have the skin prepared prior to the noraxon electrode being placed on their skin. Electrodes will be attached according to European recommendation (seniam) to the Biceps Femoris of the dominate leg. A baseline sEMG will then be taken whilst the participant is at rest for 60seconds. The electrode placement and sEMG recording will be taken by a qualified laboratory technician employed by Teesside University.

CONTACTS AND LOCATIONS:
Locations (1):
- Social Sciences, Business and Law, Middlesbrough, Teesside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chesterton P & Payton S (2017) Effects of spinal mobilisations on lumbar and hamstring ROM and sEMG: A randomised control trial. Physiotherapy Practice and Research, 38, 17-25
- [Background] Szlezak AM, Georgilopoulos P, Bullock-Saxton JE, Steele MC. The immediate effect of unilateral lumbar Z-joint mobilisation on posterior chain neurodynamics: a randomised controlled study. Man Ther. 2011 Dec;16(6):609-13. doi: 10.1016/j.math.2011.06.004. Epub 2011 Jul 13. PMID 21742541
- [Derived] Chesterton P, Evans W, Livadas N, McLaren SJ. Time-course changes associated with PA lumbar mobilizations on lumbar and hamstring range of motion: a randomized controlled crossover trial. J Man Manip Ther. 2019 May;27(2):73-82. doi: 10.1080/10669817.2018.1542558. Epub 2018 Nov 13. PMID 30935338